CLINICAL TRIAL: NCT00289081
Title: Multi-center Prospective Clinical Evaluation of the P.F.C.® Sigma™ Rotating Platform Knee Primary Cases Cruciate Retaining Versus Cruciate Substituting
Brief Title: Primary TKA Cruciate Retaining vs Cruciate Substituting With Rotating Platform Knee Prostheses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business reasons
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRP-1
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Osteoarthritis; Arthritis, Rheumatoid; Avascular Necrosis of Bone; Post-traumatic Arthritis; Rheumatoid Arthritis
Keywords: Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Rotating Platform Cruciate Retaining Knee implant
  Interventions: Device: Total Knee Replacement
- 2 (Active Comparator): Rotating Platform Cruciate Substituting Knee implant.
  Interventions: Device: Total knee replacement

INTERVENTIONS:
Device: Total Knee Replacement — Rotating Platform (RP) Cruciate Retaining Knee implant
  Other Names: P.F.C.® Sigma™ RP Cruciate Retaining Knee implant
  Arms: 1
Device: Total knee replacement — Rotating Platform (RP) Cruciate Substituting Knee implant.
  Other Names: P.F.C.® Sigma™ RP Cruciate Substituting Knee implant.
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the clinical performance of the cruciate ligament retaining or cruciate ligament substituting implants by obtaining a series of primary TKAs. Outcome scoring and radiographic assessment will be the methods used to evaluate performance.

DETAILED DESCRIPTION:
The study will evaluate the clinical performance of cruciate ligament retaining or cruciate ligament substituting implants through a series of primary TKAs. Patients will receive either the P.F.C.® Sigma™ Rotating Platform Cruciate Retaining Knee implant or the P.F.C.® Sigma™ Rotating Platform Cruciate Substituting Knee implant and assignment will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis
* Rheumatoid arthritis
* Avascular necrosis (AVN) of bone
* Other inflammatory arthritis
* Post-traumatic arthritis
* Juvenile rheumatoid arthritis

Exclusion Criteria:

* Prior ipsilateral TKA
* Metabolic disorders
* Joint replacement due to autoimmune disorders
* History of recent/active joint sepsis
* Charcot neuropathy
* Psycho-social disorders that would limit rehabilitation
* Greater than 75 years of age at the time of surgery
* Severe diabetes mellitus
* Skeletal immaturity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2001-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Knee Society scores | Pre-operative, 6 and 12 months and annually thereafter for at least 5 years.

SECONDARY OUTCOMES:
Complications | On-going to end of study
Revisions | On-going to end of study
Medical imaging | Pre-operative, 6 and 12 months and annually thereafter for at least 5 years.
SF-12 patient outcomes | Pre-operative, 6 and 12 months and annually thereafter for at least 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy L O'Dell, EMT, CCRA, Study Director — DePuy Orthopaedics
Locations (4):
- United States (4):
  - La Jolla, California
  - West Coast Orthopaedic Specialists, Crystal River, Florida
  - Melbourne, Florida
  - Cleveland Heights, Ohio